CLINICAL TRIAL: NCT03133663
Title: Heart Rate Evaluation and Resuscitation Trial in Preterm Neonates
Acronym: HEART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Vishal Kapadia, Assistant Professor of Pediatrics, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 092016-048
Record Dates: First submitted 2017-04-22; First posted 2017-04-28 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Neonatal Resuscitation; Infant, Premature
Keywords: electrocardiogram; premature; resuscitation
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Pulse oximeter and auscultation to determine heart rate during neonatal resuscitation. Pulse oximeter will be used to determine oxygen saturation.
  Interventions: Other: Pulse oximeter and auscultation group
- Electrocardiogram group (Experimental): Electrocardiogram to determine heart rate during neonatal resuscitation. Pulse oximeter will still be used per Neonatal Resuscitation Program guidelines for oxygen saturation.
  Interventions: Other: Electrocardiogram group

INTERVENTIONS:
Other: Electrocardiogram group — Experimental
  Arms: Electrocardiogram group
Other: Pulse oximeter and auscultation group — Control
  Arms: Control group

SUMMARY:
The purpose of this study is to determine whether using electrocardiograms (ECGs) during resuscitation of preterm infants (less than 31 weeks gestation) will decrease the amount of time it takes from birth for heart rate (HR) to be above 100 beats per minute and oxygen saturations to be in the goal range, in other words to stabilize the infant. A few studies have been conducted which showed that ECGs are faster at detecting HR than pulse oximetry (PO). Sample sizes, however, have been small and only few extremely low birthweight infants have been included. It is unclear if use of ECG in these tiny preterm infants in addition to traditional techniques to determine HR will be beneficial and impact resuscitation and outcomes. The investigators propose a study where infants will be randomized to either using ECG in addition to PO ± auscultation versus PO ± auscultation only to assess HR during neonatal resuscitation. The investigators hypothesize that the group of infants randomized to ECG will be able to stabilize faster, i.e. achieve HR > 100 beats per minute and oxygen saturation in goal range faster.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants less than <31 weeks gestation born at Parkland hospital vaginally or by C/S
* Infant with congenital heart disease, congenital anomalies, or chromosomal abnormalities will be included unless comfort care has been agreed upon beforehand
* Resuscitation team present to attend delivery before birth

Exclusion Criteria:

* Any infant with prenatally agreed upon comfort care since resuscitation will not be provided
* Any precipitous delivery since resuscitation team will not be in attendance prior to delivery

Max Age: 1 Hour | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
Time to Infant Stabilization | During delivery room resuscitation, up to 1 hour
  Amount of time it takes from birth for heart rate to be above 100 beats per minute and oxygen saturation to be in the goal range (per Neonatal Resuscitation Program guidelines)

SECONDARY OUTCOMES:
Time to heart rate >100 beats per minute | During delivery room resuscitation, up to 1 hour
  Time in delivery room
Time to goal oxygen saturation | During delivery room resuscitation, up to 1 hour
  Time in delivery room
Time of positive pressure ventilation | During delivery room resuscitation, up to 1 hour
  Total time positive pressure received in delivery room
Incidence of positive pressure ventilation | During delivery room resuscitation, up to 1 hour
  Positive pressure ventilation applied in delivery room
Incidence of CPR | During delivery room resuscitation, up to 1 hour
  CRP applied in delivery room
Incidence of intubation | During delivery room resuscitation, up to 1 hour
  Intubation in delivery room
Maximum FiO2 applied | During delivery room resuscitation, up to 1 hour
  FiO2 applied in delivery room
Maximum peak inspiratory pressure | During delivery room resuscitation, up to 1 hour
  Maximum peak inspiratory pressure in delivery room
Incidence of hypothermia | Until hospital discharge, up to 6 months
  Hypothermia on admission to NICU
Incidence of need for surfactant | Until hospital discharge, up to 6 months
  Surfactant given while in NICU
Incidence of bronchopulmonary dysplasia | Until hospital discharge, up to 6 months
  Incidence in NICU
Incidence of respiratory distress syndrome | Until hospital discharge, up to 6 months
  Incidence in NICU
Incidence of pneumothorax | Until hospital discharge, up to 6 months
  Incidence in NICU
Incidence of intraventricular hemorrhage | Until hospital discharge, up to 6 months
  Incidence in NICU
Incidence of necrotizing enterocolitis | Until hospital discharge, up to 6 months
  Incidence in NICU
Incidence of sepsis | Until hospital discharge, up to 6 months
  Incidence in NICU
Incidence of symptomatic PDA | Until hospital discharge, up to 6 months
  Incidence in NICU
Incidence of appropriate vs inappropriate use of positive pressure ventilation | During delivery room resuscitation, up to 1 hour
  Use in delivery room
Incidence of equipment failure of pulse oximeter and electrocardiogram | During delivery room resuscitation, up to 1 hour
  Failure in delivery room

CONTACTS AND LOCATIONS:
Locations (1):
- Parkland Hospital, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No